CLINICAL TRIAL: NCT01652170
Title: The Performance of the APPY1 Test in the Evaluation of Possible Acute Appendicitis in Children, Adolescents, and Young Adults Presenting to the Emergency Department
Brief Title: The Performance of the APPY1 Test in the Evaluation of Possible Acute Appendicitis
Acronym: APPY1
Status: Completed | Type: Observational
Sponsor: Venaxis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP12-001
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surplus plasma samples will be retrieved by the Sponsor for future development of protein biomarkers.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will consist of a brief interaction with the subject or parent or guardian to obtain consent, collect a blood sample, medical history, and physical examination of those who meet the inclusion criteria. The blood sample will be tested for the WBC value, as well as processed into plasma in order to compute the APPY1 Test result, which is based on a combination of the WBC value and the plasma MRP 8/14 and CRP concentrations received from the APPY1 Test cassette. There will be a 2-week (14 days +/- 3) follow-up telephone call for those subjects that were discharged from the ED without an appendectomy or diagnosis of acute appendicitis. Use of the APPY1 Test to help identify low risk patients could significantly reduce the use of CT scans in diagnosis of AA, thereby reducing the exposure to ionizing radiation in children, adolescents, and young adults.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 20 years old (up until the 21st birthday),
* Right lower quadrant or poorly localized abdominal pain, or tenderness that includes the right lower quadrant, and/or other features including, but not limited to, nausea, vomiting, and/or anorexia, requiring acute appendicitis to be added to the differential,
* Onset of abdominal pain within 72 hours or less,
* Patients of either gender may participate and,
* Patient or accompanying parent or guardian is able to provide informed consent.

Exclusion Criteria:

* History includes prior appendectomy,
* Subjects whose presentation history and physical examination place them at such high risk of acute appendicitis that it would be clinically reasonable to proceed with exploratory laparotomy and/or appendectomy without advanced imaging,
* Treatment with any immunosuppressive medication or chemotherapeutic agents within 28 days, or systemic steroids (oral or intravenous) within 14 days,
* History of end-stage, metastatic cancer or an active immune disorder,
* History includes abdominal trauma or invasive abdominal procedures/surgery within the previous two weeks,
* Patients who have received diagnostic imaging (CT, MRI, or US) for abdominal pain in the previous two weeks,
* Patients with report of abdominal pain greater than 72 hours,
* History of active bleeding disorder, which may complicate phlebotomy or placement of peripheral IV catheter,
* Participation in a research study within the previous 30 days,
* Prisoners of an adult or juvenile detention center, and
* Subject, parent or guardian unable to provide informed consent.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults 2 to 20 years old.
Sampling Method: Non-Probability Sample
Enrollment: 2201 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity, Specificity, Negative and Positive Predictive Value | Upon 3rd party review of data
  95% confidence intervals on Sensitivity and Specificity

SECONDARY OUTCOMES:
CT utilization | Upon 3rd party review of data
  CT utilization behaviors based on questions posed to the physicians about their current imaging intentions and those intentions were an APPY1 Test result available

CONTACTS AND LOCATIONS:
Overall Officials: Dave Huckins, MD, Principal Investigator — Newton-Wellesley Hospital
Locations (29):
- United States (29):
  - Phoenix Children's Hosptial, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC Davis, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, College of Medicine, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Emory-Egleston (CHOA), Atlanta, Georgia
  - Scottish Rite (CHOA), Atlanta, Georgia
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - University of Michigan, Mott Children's Hospital, Ann Arbor, Michigan
  - Spectrum Health System, Grand Rapids, Michigan
  - The Children's Mercy Hosptial, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Staten Island University Hospital, Staten Island, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's, Columbus, Ohio
  - OHSU, Portland, Oregon
  - Children's Hospital of Pittsburg, Pittsburgh, Pennsylvania
  - Rhode Island Hospital - Hasbro, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - St. Joseph's Regional Health Center, Bryan, Texas
  - St. Joseph's Emergency Center, College Station, Texas
  - Dallas Children's Hospital, Dallas, Texas